CLINICAL TRIAL: NCT04431843
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Spirulina Maxima Extract on Improvement of Cognitive Function
Brief Title: the Efficacy and Safety of Spirulina Maxima Extract on Improvement of Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KIOST-CF-SM2
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Function
Keywords: Spirulina maxima Extract; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina maxima extract (Experimental): Spirulina maxima extract for 1.5 g/day
  Interventions: Dietary Supplement: Spirulina maxima extract
- Placebo (Placebo Comparator): Spirulina maxima extract for 0 g/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Spirulina maxima extract — once a day for 2 p.o., after breakfast and dinner(1.52 g/day, Spirulina maxima extract for 1.5 g/day) for 12 week
  Arms: Spirulina maxima extract
Dietary Supplement: Placebo — once a day for 2 p.o., after breakfast and dinner(1.52 g/day, Spirulina maxima extract for 0 g/day) for 12 week
  Arms: Placebo

SUMMARY:
This study was the evaluate the efficacy and safety of Spirulina maxima extract on the improvement of Cognitive Function

DETAILED DESCRIPTION:
This study was 12 weeks, randomized, double-blind, placebo-controlled human trial to evaluate. 80 subjects participated in Spirulina maxima extract or placebo group. To evaluate the changes in the evaluation items when Spirulina maxima extract was taken 12 weeks compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are at least 60 years of age at screening
* Persons who have Korean Mini-Mental Status Examination(K-MMSE) result in 25-28 points
* Persons who agree to voluntary participation and to comply with the Notice after fully hearing and understanding the details of this human trial

Exclusion Criteria:

* Patients with a past history of treatment with Axis I disorder in SCID(Structured Clinical Interview for DSM-IV) which is a structured clinical interview in the Diagnostic and Statistical Manual of Mental Disorders at Screening or who have been treated within the last 3 years
* Patients with BMI(Body Mass Index)<18.5 kg/m^ or 35 kg/m^≤BMI(Body Mass Index)
* Patients with alcohol abuse or dependence within the last 3 months
* Patients who have clinically significant following severe illness (i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.)
* Patients with a history of clinically significant hypersensitivity to Spirulina Maxima
* Patients taking medicines, health functional foods or herbal medicines related to the improvement of cognitive function and memory within 1 month before screening
* Patients who ingested Spirulina Maxima extract's health functional food within 1 month before screening
* Patients who whole blood donation within 1 months before the first ingestion or Component blood donation within 2 weeks
* Patients who participate in another human trial within 3 months
* Those who show the following results in the Laboratory test

  * AST, ALT > 3 times upper limit of the normal range
  * Other significant laboratory test opinion
* Patients who are deemed unsuitable for participating in the human trial due to other reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Changes of Visual learning test | 12 weeks
  Visual learning test of CNT(Computerized neurocognitive function test) was measured in baseline and 12 week. And changes of result from the test were utilized.
Changes of Visual working memory test | 12 weeks
  Visual working memory test of WMT(working memory tasks) was measured in baseline and 12 week. And changes of result from the test were utilized.
Changes of Verbal learning test | 12 weeks
  Verbal learning test of CNT(Computerized neurocognitive function test) was measured in baseline and 12 week. And changes of result from the test were utilized.

SECONDARY OUTCOMES:
MoCA-K; Korean Version of the Montreal Cognitive Assessment | 12 weeks
  The cognitive function evaluation using the Montreal Cognitive Assessment(MoCA-K) is a total of 8 items, and evaluates cognitive functions such as time / execution power, vocabulary, memory, attention, sentence, abstraction, delayed recall, and orientation.
  Time / execution power's total score is 5 points, vocabulary's total score is 3 points, attention's total score is 3 points, sentence's total score is 3 points, abstraction's total score is 2 points, delayed recall's total score is 5 points, orientation's total score is 6 points. It takes about 10 minutes to complete, and the total score is 30 points and total score make sum score. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.
  It takes about 10 minutes to complete, and the score is 30 points. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.
Changes of Auditory continuous performance test | 12 weeks
  Auditory continuous performance test of CNT(Computerized neurocognitive function test) was measured in baseline and 12 week. And changes of result from the test were utilized.
BDNF; Brain-derived neurotrophic factor | 12 weeks
  Brain-derived neurotrophic factor(BDNF)(pg/mL) was measured in baseline and 12 week.
Changes of TAS(Total antioxidant status) | 12 weeks
  Total antioxidant status(TAS) was measured in baseline and 12 week. And changes of result from the test were utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Department of Psychiatry, Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea